CLINICAL TRIAL: NCT01884168
Title: Gene Expression Profiling and Immunological Mechanism Affects the Response of Malignant Cavity Effusion Towards DC-CIK Immunotherapy
Brief Title: Study of Gene Expression Profiling and Immunological Mechanism Affects the Response of Immunotherapy
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Director, Capital Medical University
Other Study IDs: GIMCEI
Record Dates: First submitted 2013-06-19; First posted 2013-06-21 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- gene expression profile: T-Cell Receptor/B-Cell Receptor gene expression in cavity effusion is detected by micro-array to explore the mechanism that DC-CIK immunotherapy controls the malignant cavity effusion.
  Interventions: Biological: Dc-CIK immunotherapy

INTERVENTIONS:
Biological: Dc-CIK immunotherapy — The patients with malignant cavity effusion are treated with dendritic cells (DC) plus cytokine induced killer cells (CIK) locally.

SUMMARY:
To investigate gene expression profile and immunological associated analysis relating to immunotherapy response of patients with malignant tumor presenting malignant cavity effusion after DC-CIK immunotherapy.

DETAILED DESCRIPTION:
1. The patients with malignant cavity effusion are treated with dendritic cells (DC) plus cytokine induced killer cells (CIK) locally.
2. Malignant cavity effusion from cancer patients is obtained through puncture and is centrifugalized to get supernatant fluid and enrich cancer cells before and after the therapy.
3. The enriched cancer cells which are flash frozen, as well as the supernatant, are stored at -80°C until processing.
4. The T-Cell Receptor/B-Cell Receptor gene expression in cavity effusion is detected by micro-array to explore the mechanism that DC-CIK immunotherapy controls the malignant cavity effusion.
5. Statistical analysis is performed using unsupervised hierarchical cluster.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed with malignant tumor and malignant cavity effusion.
2. An Eastern Cooperative Oncology Group（ECOG）performance status of 0-2.
3. Normal cardiac, hepatic, renal and bone marrow functions.
4. Life expectancy >3 months.
5. Not receive other anti-tumor treatment.
6. Not receive chemotherapy in pleural and abdominal cavity.

Exclusion Criteria:

1. Previous history of other malignancies.
2. Serious or uncontrolled concurrent medical illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The malignant tumor patients present with malignant cavity effusion and can receive DC-CIK immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2022-12 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Immunotherapy response | 1 month
  T-Cell Receptor and B-Cell Receptor gene expression profiling and the change of cytokines, lymphocytes subpopulation before and after DC-CIK infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ren, MD, PhD, Principal Investigator — Capital Medical University Cancer Center /Beijing Shijitan Hospital
Locations (1):
- Capital Medical University Cancer Center/Beijing Shijitan Hospital, Beijing, Beijing Municipality, China